CLINICAL TRIAL: NCT07228897
Title: Evaluation of the Effect of Open-Air Walking Supported by Treadmill and Mobile Application on Cardiopulmonary Function and Quality of Life in Patients With Fibromyalgia Syndrome
Brief Title: Comparison of Treadmill and Outdoor Walking in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-182
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open air walking (Experimental)
  Interventions: Other: Walking exercises at open air place
- treadmill (Active Comparator)
  Interventions: Other: Walking exercises with treadmill

INTERVENTIONS:
Other: Walking exercises with treadmill — Patients will be enrolled in a treadmill exercise program in the cardiopulmonary exercise unit for 45 minutes, 3 days a week for 4 weeks.
  Arms: treadmill
Other: Walking exercises at open air place — Patients will walk briskly outdoors for 45 minutes, 3 days a week for 4 weeks. Patients will receive notifications via a mobile app reminding them of their daily walk, and they will be asked to log their walks in the mobile app.
  Arms: Open air walking

SUMMARY:
While walking exercises performed outdoors are important within the scope of aerobic exercise, the continuity of outdoor walking exercises can be negatively affected by different weather conditions. Walking exercises performed indoors on a treadmill are a good option for patients in terms of increasing exercise continuity and patient compliance. Walking outdoors supported by a treadmill and mobile application may increase aerobic capacity and quality of life in patients with fibromyalgia syndrome, as well as reduce kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 25 and 55
2. Be female
3. Have not engaged in regular physical activity for the past 3 months
4. Have been using the same medical treatment for at least 1 month prior to the study (amitriptyline, duloxetine/milnacipran, pregabalin, cyclobenzaprine)
5. Volunteering to participate in the study
6. The patient's cognitive status being suitable for using a mobile application
7. The patient agreeing to the 'Personal Data Protection Law Information Text' in order to use the mobile application

Exclusion Criteria:

1. History of cardiac or pulmonary disease
2. Changes in medical treatment during the study period
3. Use of different injection methods (ozone therapy, neural therapy, acupuncture, etc.) at least 3 months prior to the study or during the study period
4. History of rheumatological disease
5. Pregnancy or breastfeeding
6. History of malignancy
7. Presence of psychiatric or neurological disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | First day of treatment, at the end of 4 week

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | First day of treatment, at the end of 4 week
Measurement of maximum inspiratory and expiratory pressure (MIP) and (MEP) | First day of treatment, at the end of 4 week
Beck Depression Scale | First day of treatment, at the end of 4 week
Fatigue Impact Scale | First day of treatment, at the end of 4 week
Short Form-36 (SF-36) | First day of treatment, at the end of 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)